CLINICAL TRIAL: NCT05475834
Title: A Phase I Study to Investigate The Mass Balance and Biotransformation of SIM0417 in Healthy Adult Chinese Male Participants
Brief Title: Study to Investigate the Mass Balance and Biotransformation of SIM0417 in Healthy Adult Chinese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM0417-104
Record Dates: First submitted 2022-07-20; First posted 2022-07-27 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Healthy Male Volunteers
Keywords: Mass Balance
MeSH Terms: interventions — SIM0417

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIM0417 (Experimental): Single oral dose of 750 mg SIM0417 coadministered with 100 mg ritonavir.
  Interventions: Drug: SIM0417

INTERVENTIONS:
Drug: SIM0417 — Single oral dose of 750 mg SIM0417 coadministered with 100 mg ritonavir.

SUMMARY:
This is a non-randomized, open-label, single-dose, Phase I clinical study to evaluate the mass balance and biotransformation, safety and tolerability of SIM0417 in healthy Chinese adult male subjects following a single oral administration of SIM0417 in combination with ritonavir.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, open-label, single-cohort, single-dose, Phase I clinical study to evaluate the mass balance, biotransformation, safety, and tolerability of SIM0417 following a single oral administration of SIM0417 combination with ritonavir in healthy Chinese adult male subjects.

This study is planned to enroll 6-8 healthy male subjects, each subject will receive SIM0417 combined with ritonavir administration. SIM0417 is single dosed, and ritonavir is administered 12 hours before SIM0417 administration (-12h), at the time of SIM0417 administration (0h), 12h (12h), and 24h (24h) after SIM0417 administration.

SIM0417 is administered after meals, ritonavir is administered either in fasting condition or after meals.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the research content, process, and potential risks of this trial, voluntarily participate in the clinical trial and sign the informed consent.
2. Healthy male subjects aged ≥18 years and ≤55 years old.
3. Body weight ≥50 kg, body mass index ≥19 kg/m2 and ≤28 kg/m2.
4. Subjects agree to take recognized effective contraceptive measures during the study period and within 3 months after the last dose of the study drug, starting from signing the informed consent.

Exclusion Criteria:

1. Any diseases that may affect the study results or the safety and status of the subjects, including but not limited to the central nervous system, respiratory system, cardiovascular system, alimentary system, blood and lymphatic system, endocrine system, musculoskeletal system, hepatic and kidney function obstacle.
2. Difficulty in venous blood collection, a history of fainting blood or needles, or those who cannot tolerate blood collection with intravenous indwelling needles.
3. With dysphagia or any history of gastrointestinal diseases that affect drug absorption/metabolism/excretion (including habitual constipation or diarrhea, perianal disease or hematochezia, irritable bowel syndrome, inflammatory bowel disease, etc.).
4. Have special requirements for diet and cannot comply with the provided diet and corresponding regulations.
5. With specific allergic history ( asthma, urticaria, eczema, etc. ) or allergic constitution ( such as those allergic to two or more drugs, food such as milk, and pollen ) are allergic to any component of the research drug or research drug.
6. Have taken special diet ( including of pitaya, mango, grapefruit, food or beverage containing caffeine, etc. ) or intense exercise within 48 h before the first administration of the drug.
7. Any prescription, non-prescription, vitamin, or herbal medicine was taken within 4 weeks before and during the screening period.
8. During the first 3 months prior to screening or from the screening period to the first administration period, alcohol was often consumed, i.e., more than 2 units of alcohol per day ( 1 unit = 360 mL beer or 45 mL spirits with 40 % alcohol or 150 mL wine ); or alcohol breath test positive.
9. More than 5 cigarettes per day during the 3 months prior to screening.
10. Participated in any drug clinical trial as a subject within 3 months prior to screening and took the study drug.
11. With blood donation or blood loss was greater than 200 mL within 3 months prior to screening, or blood transfusion or blood products were received within 4 weeks.
12. Have a history of drug abuse or be positive in drug abuse screening test.
13. At the time of screening, the blood pressure in the resting state and the pulse are within the following ranges: such as systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg, pulse <55 bpm or >100 bpm.
14. Electrocardiographic QTc > 450 msec (Fridericia formula) at screening, or presence of risk factors for Torsade de Pointes (eg, history of heart failure, history of hypokalemia, family with prolonged QT syndrome) history), or other abnormal clinical significance (judged by the investigator).
15. HBV surface antigen, HCV antibody, HIV, or syphilis are positive during screening.
16. Physical examination, vital signs, blood routine, blood biochemistry ( serum creatinine > 1.0 × ULN )), coagulation function, thyroid function, urine examination, chest X-ray, abdominal B-scan ultrasonography, thyroid B-scan ultrasonography results were abnormal and have clinical significance (judged by the investigator).
17. Those who have been vaccinated within 1 month before screening (except for the novel coronavirus vaccine), or who plan to be vaccinated during treatment / within 2 weeks after the last dose of study drug.
18. Be positive in SARS-CoV-2 nucleic acid test at screening.
19. Subjects have other conditions that are not suitable for participating in this research, or the subjects may not be able to complete this research for other reasons (judged by the investigator).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
Total recovery of SIM0417-related substances in urine | Up to 168 hours(approx) from SIM0417 administration
  Total recovery of SIM0417-related substances in urine after a single dose of SIM0417 in combination with ritonavir, elucidating the main route of excretion, and clarifying the cumulative recovery of the parent drug and its metabolites (if applicable)
Total recovery of SIM0417-related substances in feces | Up to 168 hours(approx) from SIM0417 administration
  Total recovery of SIM0417-related substances in feces after a single dose of SIM0417 in combination with ritonavir, elucidating the main route of excretion, and clarifying the cumulative recovery of the parent drug and its metabolites (if applicable)
Identification of metabolites in plasma | Up to 72 hours (approx) from SIM0417 administration
  Identification of metabolites in plasma (if applicable), to identification of major biotransformation pathways
Identification of metabolites in urine | Up to 168 hours (approx) from SIM0417 administration
  Identification of metabolites in urine (if applicable), to identification of major biotransformation pathways
Identification of metabolites in feces | Up to 168 hours (approx) from SIM0417 administration
  Identification of metabolites in feces (if applicable), to identification of major biotransformation pathways

SECONDARY OUTCOMES:
Adverse Events | Up to 14 days from SIM0417 administration
  Number of Participants With Adverse Events
Vital Signs | Up to 8 days from SIM0417 administration
  Number of Participants With Clinically Notable Vital Signs
ECG | Up to 8 days from SIM0417 administration
  Number of Participants With Clinically Notable Electrocardiogram (ECG) Values
Laboratory Tests | Up to 8 days from SIM0417 administration
  Number of Participants With Clinically Notable Laboratory Tests

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Shandong First Medical University
Locations (1):
- Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No